CLINICAL TRIAL: NCT05494385
Title: Effect of Perioperative Gabapentin on Postoperative Opioid Requirements
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglass Hale, Adjunct Clinical Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBGYN-IIR-PERI-OP-GABAPENTIN
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Gabapentin/Postoperative Placebo (Placebo Comparator)
  Interventions: Drug: Preoperative Gabapentin/Postoperative Placebo
- Preoperative Gabapentin/Postoperative Gabapentin (Active Comparator)
  Interventions: Drug: Preoperative Gabapentin/Postoperative Gabapentin

INTERVENTIONS:
Drug: Preoperative Gabapentin/Postoperative Placebo — Postoperatively, this group will receive scheduled acetaminophen and ibuprofen every 6 hours, in addition to placebo every 12 hours. The placebo is encapsulated to appear identical to the active drug. This group will have oxycodone 5 mg every 6 hours as needed for pain.
  Arms: Preoperative Gabapentin/Postoperative Placebo
Drug: Preoperative Gabapentin/Postoperative Gabapentin — Postoperatively, this group will receive scheduled acetaminophen and ibuprofen every 6 hours, in addition to gabapentin every 12 hours. The gabapentin is encapsulated to appear identical to the placebo. This group will have oxycodone 5 mg every 6 hours as needed for pain.
  Arms: Preoperative Gabapentin/Postoperative Gabapentin

SUMMARY:
The purpose of this study is to determine if preoperative gabapentin is noninferior to preoperative and postoperative gabapentin for pain control in patients undergoing surgery for pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years old
* English-speaking
* Stage > 2 pelvic organ prolapse
* Undergoing pelvic organ prolapse procedure (including native tissue vaginal procedure, native tissue laparoscopic procedure, mesh-augmented laparoscopic procedure, obliterative procedure)
* Planning overnight stay

Exclusion Criteria:

* Renal dysfunction (creatinine clearance <60 mL/min)
* Allergy to acetaminophen and ibuprofen
* Allergy to gabapentin
* Patients on a Controlled Substance Agreement or Opioid Contract from another provider. This information is available in the IU Health electronic medical record, Cerner.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglass S Hale, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Started | 59 | 55
Completed | 59 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin | Total
Number analyzed (Participants) | 59 | 55 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (11.1) | 59.8 (12.9) | 59.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 55 | 114
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 54 | 49 | 103
  Non-Hispanic Black | 3 | 3 | 6
  Hispanic or Latino | 2 | 2 | 4
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Opioid Prescription at Discharge
Description: Percentage of patients requiring an opioid prescription at discharge in each group. Patients who use 5 or more doses of PRN opioids during inpatient postoperative course will receive a prescription for opioids.
Time Frame: Length of postoperative hospital stay (at discharge, an average of 32 hours from time of registration for surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
Participants
  Opioid prescription at discharge | 40 | 40
  No opioid prescription at discharge | 19 | 15

2. Secondary Outcome: Opioid Refill Requests
Description: Number of patients in each group who call the office to request a new opioid prescription (if they were discharged without a prescription) or to request an opioid prescription refill (if they were discharged with a prescription) within the 6-week postoperative time period.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
Participants
  Refill/new opioid prescription within 6 weeks | 50 | 49
  No refill/new opioid prescription within 6 weeks | 9 | 6

3. Secondary Outcome: Inpatient Pain Scores
Description: Pain scores in the hospital will be measured on a numeric rating scale (0-10) with 0 being no pain and 10 being worst pain. Highest pain score recorded.
Time Frame: Length of postoperative hospital stay (an average of 32 hours following surgery)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
units on a scale | 6 [5 to 8] | 7 [4 to 8]

4. Secondary Outcome: Inpatient Morphine Milligram Equivalents
Description: Total morphine milligram equivalents used will be calculated by converting total PO and IV opioids used postoperatively until hospital discharge to morphine milligram equivalents using the opioid equianalgesic chart.
Time Frame: Length of postoperative hospital stay (an average of 32 hours following surgery)
Measure: Median (Full Range); unit: morphine milligram equivalenst
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
morphine milligram equivalenst | 15 [0 to 30] | 7.5 [0 to 22.5]

5. Secondary Outcome: Length of Stay
Description: Length of stay will be measured in hours by time of registration for surgery to time of discharge from hospital.
Time Frame: Time of registration for surgery to time of discharge from hospital
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
hours | 32.8 (7.6) | 31.0 (4.3)

6. Secondary Outcome: Nausea
Description: Nausea will be measured by the number of "as needed" antiemetics the patient received postoperatively.
Time Frame: Length of postoperative hospital stay (an average of 32 hours following surgery)
Measure: Median (Full Range); unit: antiemetics used
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 59 | 55
antiemetics used | 0 [0 to 1] | 0 [0 to 1]

7. Secondary Outcome: Sedation
Description: Sedation will be measured by the Stanford Sleepiness Scale. This is a self-administered scale that the patient will complete at 10AM on postoperative day 1.
Time Frame: On postoperative day 1 between 6AM and 10AM
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
Number analyzed (Participants) | 48 | 50
Participants
  Feeling active, vital, alert, or wide awake | 13 | 15
  Functioning at high levels, but not at peak; able to concentrate | 19 | 15
  Awake, but relaxed; responsive but not fully alert | 8 | 12
  Somewhat foggy, let down | 5 | 3
  Foggy; losing interest in remaining awake; slowed down | 2 | 1
  Sleep, woozy, fighting sleep; prefer to lie down | 1 | 4
  No longer fight sleep, sleep onset soon, having dream-like thoughts | 0 | 0

ADVERSE EVENTS:
Time Frame: Each participant was assessed from time of surgery until their six week postoperative visit, an average of 6 weeks.
Arm/Group | Preoperative Gabapentin/Postoperative Placebo | Preoperative Gabapentin/Postoperative Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/55
Other Adverse Events (participants affected / at risk) | 0/59 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05494385/Prot_SAP_001.pdf